CLINICAL TRIAL: NCT04606550
Title: Randomized Clinical Trial Comparing the MonaLisa Laser Versus Vaginal Estrogen in Post-Menopausal Breast Cancer Patients: a SHE CAN Non-inferiority Study
Brief Title: MonaLisa Laser Intervention for Post-Menopausal Breast Cancer Patients: A SHE CAN Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No financial support.
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Christine Brezden-Masley, Principal Investigator, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-0140-A
Record Dates: First submitted 2020-10-09; First posted 2020-10-28 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer Female; Genitourinary Syndrome of Menopause

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vaginal Laser HR+ (Experimental): During our study, women will undergo treatment intravaginally and vulvar with the fractional microablative CO2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy). A treatment cycle includes three laser applications (every 40-50 days, approximately 6 weeks). The procedure will be performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia).
  Interventions: Device: Microablative Fractional CO2 Laser Therapy
- Vaginal Estrogen HR- (Active Comparator): The women in the vaginal estrogen group will be prescribed and asked to administer: Conjugated estrogen cream (Premarin®): 0.5 g of cream intravaginally daily (using applicator or fingertip) for two weeks (fourteen days) then 0.5 g twice weekly for 24 ± 2 additional weeks.
  Interventions: Device: Microablative Fractional CO2 Laser Therapy
- Vaginal Laser HR- (Active Comparator): During our study, women will undergo treatment intravaginally and vulvar with the fractional microablative CO2 laser system (SmartXide 2 V 2 LR, MonaLisa Touch, DEKA, Florence, Italy). A treatment cycle includes three laser applications (every 40-50 days, approximately 6 weeks). The procedure will be performed in the outpatient clinic and does not require any specific preparation (e.g. analgesia/anesthesia).
  Interventions: Device: Microablative Fractional CO2 Laser Therapy

INTERVENTIONS:
Device: Microablative Fractional CO2 Laser Therapy — Microablative Fractional CO2 Vaginal Laser Therapy
  Other Names: MonaLisa Laser

SUMMARY:
The purpose of this study is to assess the efficacy of a fractional CO2 laser ("SmartXide2 - V2LR", DEKA M.E.L.A., Florence - Italy) "the Laser" in the treatment of genitourinary symptoms of menopause, female sexual function, and urogenital health in comparison to vaginal estrogen. Only breast cancer patients who have HR (-) breast cancer are planning to be included in the vaginal estrogen group.

DETAILED DESCRIPTION:
The investigators aim to determine the efficacy of the MonaLisaTouch Laser in comparison with vaginal estrogen in the management and treatment of GSM symptoms resulting in vaginal atrophy, sexual dysfunction and a decreased quality of life in women with a history of breast cancer. Patients will be stratified according to menopausal status prior to breast cancer therapy and HR tumor status. Fractional CO2 laser therapy has been approved by Health Canada for use in menopausal women with GSM, nevertheless long term efficacy and safety data is lacking in the breast cancer survivor population. In the short term (i.e. 6 month follow up), research has shown that this therapy is a safe and effective treatment that has promising benefits with little to no reported adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written and voluntary informed consent understood, signed and dated
2. Aged between 18 and 75 years old
3. Have had previous histologically-proven diagnosis of breast cancer
4. Have moderate to severe GSM symptoms as determined by their treating oncologist or another responsible physician.
5. Interested in receiving treatment for their GSM symptoms, and willing to be randomized to a treatment arm in this protocol.
6. Completed chemotherapy and / or radiation treatment at least 3 months prior to starting the study, and/or maintenance endocrine therapy for at least 3 months prior to starting the study.
7. For hormone receptor negative cohort, must be post-menopausal
8. ECOG status <2

Exclusion Criteria:

1. Have a suspected or diagnosed gynecological illness or malignancy.
2. Inability to attend outpatient clinics for any reason.
3. Inability to provide consent or complete the questionnaire (e.g. Language barrier, concerns about competence)
4. Contraindication to vaginal estrogen therapy
5. Personal history of thrombophlebitis, heart failure, or myocardial infarction within 12 months, scleroderma, or any chronic condition that could interfere with study compliance.
6. Pelvic organ prolapse higher than stage II, pelvic surgery within 6 months, or previous reconstructive pelvic surgery with transvaginal mesh kits.
7. Have used vaginal estrogen cream, ring or tablet within 1month before entering the study, or vaginal moisturizers, lubricants or homeopathic preparations within 2 weeks of therapy.
8. Personal history of vulvovaginal condyloma, vaginal intraepithelial neoplasia (VAIN), vaginal carcinoma, lichen sclerosis, lichen planus, history of vaginal radiation, history of cervical cancer, other gynaecologic cancer, pelvic or vaginal radiation
9. Acute or recurrent urinary tract infection (UTI), or genital infection (e.g. bacterial vaginosis, herpes genitalis, candida, pelvic inflammatory disease)
10. Personal history of impaired wound healing or Scleroderma
11. History of keloid formation
12. Use or anticipated use of antiplatelet therapy, anticoagulants, thrombolytics, vitamin E or nonsteroidal anti-inflammatory drugs within 2 weeks pre-treatment

    -

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
MonaLisa Touch Impact on vaginal health in breast caner patients | 2 years
  The aim of our research, is to assess the impact of the MonaLisa Touch Laser on the sexual health and quality of life of breast cancer survivors with GSM in comparison to vaginal estrogen.
VAS | 6 months
  To compare subjective improvement of vaginal dryness in breast cancer survivors, using the 10 cm visual analog scale (VAS) for GSM symptoms 6 months post-treatment between groups.

IPD SHARING:
Plan to Share IPD: Undecided